CLINICAL TRIAL: NCT06845046
Title: A Randomized Trial to Optimize Skeletal Muscle While Reducing Adiposity in Veterans With HIV
Brief Title: A Study to Improve Skeletal Muscle in Veterans With HIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: INFA-009-24F
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: HIV; Obesity
Keywords: HIV; obesity; skeletal muscle; dietary supplement
MeSH Terms: conditions — Obesity | interventions — Carnitine

STUDY DESIGN:
Intervention Model Description: Randomization to one of 4 groups: Diet control group, Diet + w-3 supplement, Diet + L-carnitine supplement, Diet + w-3 + l-carnitine, followed by addition of resistance exercise training in each group, total intervention period is 4 weeks
Who Masked: Investigator
Masking Description: PI blinded to randomization group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control Diet (Placebo Comparator): Diet high in unsaturated fat
  Interventions: Other: Control Diet
- Diet + w-3 fatty acids (Experimental): Diet high in unsaturated fat plus omega-3 fatty acid supplement
  Interventions: Dietary Supplement: w-3 fatty acid; Other: Control Diet
- Diet + L-Carnitine (Experimental): Diet high in unsaturated fat plus L-carnitine supplement
  Interventions: Dietary Supplement: L-carnitine; Other: Control Diet
- Diet + w-3 fatty acids + L-carnitine (Experimental): Diet high in unsaturated fat plus omega-3 fatty acid supplement plus L-carnitine supplement
  Interventions: Dietary Supplement: w-3 fatty acid; Dietary Supplement: L-carnitine; Other: Control Diet

INTERVENTIONS:
Dietary Supplement: w-3 fatty acid — omega-3 fatty acid supplement
  Arms: Diet + w-3 fatty acids; Diet + w-3 fatty acids + L-carnitine
Dietary Supplement: L-carnitine — L-carnitine supplement
  Arms: Diet + L-Carnitine; Diet + w-3 fatty acids + L-carnitine
Other: Control Diet — Control Diet high in unsaturated fat

SUMMARY:
The Department of Veterans Affairs is the largest single provider of medical care to people with HIV in the United States. The condition of excess lipid within and around muscle, termed myosteatosis, predisposes Veterans to physical function decline, frailty, disability, and cardiometabolic diseases such as diabetes and cardiovascular disease. In the investigators current Merit supported cohort, the investigators found that 36% of Veterans with treated HIV and obesity have "myosteatotic type obesity". Based on the investigators findings, the investigators have designed a multipronged integrated intervention that combines: 1) dietary replacement of saturated with unsaturated fats; 2) administration of L-carnitine and omega-3 fatty acid supplementation; and 3) targeted resistance exercise training.

DETAILED DESCRIPTION:
The Department of Veterans Affairs is the largest single provider of medical care to people with HIV in the United States. With the advances achieved in antiretroviral therapy (ART), Veterans with HIV now survive decades. However, this success is tempered by the rising burden of obesity now affecting 78% of Veterans. Defects in adipose tissue lipid storage and regulation are hallmarks of both treated HIV and obesity, which leads to a high degree of ectopic fat infiltrating organs and tissues such as skeletal muscle. The condition of excess lipid within and around muscle, termed myosteatosis, predisposes Veterans to physical function decline, frailty, disability, and cardiometabolic diseases such as diabetes and cardiovascular disease. In the investigators current Merit supported cohort, the investigators found that 36% of Veterans with treated HIV and obesity have "myosteatotic type obesity". Further, the investigators found that high ectopic fat accumulation in muscle (quantified by CT imaging of skeletal muscle density) is associated with reduced mitochondrial oxidative capacity, greater inflammation, and impaired muscle glucose tolerance and insulin sensitivity. Hence the quality of muscle is just as important as the quantity of muscle. However, this important phenomenon has received little attention, especially in Veterans with HIV. Indeed, the need to target mobilizing and metabolizing skeletal muscle ectopic fat while preserving/increasing the total amount of skeletal muscle is most often overlooked and represents a major research gap and unmet clinical need. From the investigators current Merit Award funded study, the investigators have an established collaboration of experienced VA researchers with expertise in HIV and immunology, human nutrition and metabolism, endocrinology, radiology and imaging science, and muscle physiology. Based on the investigators findings, the investigators have designed a multipronged integrated intervention that combines: 1) dietary replacement of saturated with unsaturated fats; 2) administration of L-carnitine and omega-3 fatty acid supplementation; and 3) targeted resistance exercise training. This evidence-based intervention is designed to: a) increase lipid flux by facilitating the transfer of long-chain fatty acids into muscle mitochondria for -oxidation; b) decrease muscle proteolysis; and c) lessen insulin resistance and inflammation. Using a mixed 2x4 factorial design trial design in a cohort of 60 Veterans who have HIV and obesity, this study will determine the main and interaction effects of the multi-pronged intervention on: skeletal muscle density, mitochondrial oxidative capacity, and fatty acid oxidation (Aim 1); glucose tolerance, insulin sensitivity, and inflammation (Aim 2); and cardiopulmonary exercise tolerance and physical function (Aim 3). Obesity in Veterans with treated HIV is a heterogeneous condition. The investigators current Merit research shows myosteatotic obesity is a distinct condition from visceral or steatotic or sarcopenic obesity, affected by different clinical factors. The investigators findings to date provide the foundation for a novel evidence-based intervention that has the potential for significant clinical impact on Veterans, including and beyond those with HIV. This proposal meets VA-ORD priorities to improve health behaviors, focus on underserved Veterans, and provide precision care.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* HIV+
* antiretroviral therapy = integrase strand transfer inhibitor for at least 3 months
* HIV-1 RNA <50 copies/ml
* age = 20 yrs
* BMI 28-50 kg/m2

Exclusion Criteria:

* unstable body weight (gain or loss > 5% over past 3 months)
* diagnosed mitochondrial disorder
* diagnosed type 1 or type 2 diabetes
* use of metformin or other anti-diabetic agents for pre-diabetes
* hemoglobin A1c of >6.5% at screening visit
* inflammatory conditions or chronic corticosteroid use
* stage 3 or greater kidney disease
* dietary or herbal supplements known to affect body weight, muscle mass, or immune function
* MRI incompatibility
* inability to perform physical function tests due to anatomical limitations
* contradictions to CPET such as exercise-induced ischemia or supplemental oxygen

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2029-06-29 (Estimated); Study Completion 2029-06-29 (Estimated)

PRIMARY OUTCOMES:
Myosteatosis | Week 24 and 44
  CT quantified abdominal skeletal muscle density
MixedMeal GTT | Week 24 and 44
  IV Glucose tolerance testing after consumption of BOOST as a meal substitute
Physical Function | Week 24 and 44
  Physical Function Testing using Hand Grip Strength Dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Heidi J Silver, PhD, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN; John R Koethe, MD, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (1):
- Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No